CLINICAL TRIAL: NCT03664271
Title: Randomized Controlled Trial of an Educational Eczema Video
Brief Title: Educational Eczema Video Intervention
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Corinna Rea, Assistant in Medicine, Principal Investigator, Instructor in Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P00029896
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Eczema
Keywords: atopic dermatitis; eczema
MeSH Terms: conditions — Eczema; Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- in-clinic video intervention (Experimental): Intervention: Caregivers will watch an educational video in clinic, and also be given information about how to access the video from home (ideal condition). The intervention video will contain educational information about eczema, as well as routine skincare and common treatments.
  Interventions: Behavioral: in-clinic video intervention
- at home video intervention (Active Comparator): Intervention: Caregivers will be given information about how to watch the video at home, but will not watch it in clinic (real-world condition).The intervention video will contain educational information about eczema, as well as routine skincare and common treatments.
  Interventions: Behavioral: at home video intervention
- usual care (No Intervention): Control: Caregivers will not watch the educational video, but will be given access to it at the conclusion of the study.

INTERVENTIONS:
Behavioral: in-clinic video intervention — Video with information about eczema and eczema treatment, to be watched in clinic and at home
  Arms: in-clinic video intervention
Behavioral: at home video intervention — Video with information about eczema and eczema treatment, to be watched at home only
  Arms: at home video intervention

SUMMARY:
The objectives of this study are to increase families' understanding of eczema and improve eczema management in the primary care setting. The investigators plan to create an educational video for families providing general information about eczema as well as instructions about good skincare management and common treatments. The investigators will conduct a randomized controlled trial of the plan in the primary care clinic at Boston Children's Hospital. Specifically, the investigators aim to (1) decrease eczema severity (2) improve patient and family quality of life (QOL) and (3) increase parental knowledge about eczema and eczema management.

ELIGIBILITY:
Inclusion Criteria:Eligibility criteria include the following:

* accompanying adult speaks English
* patient has a history of eczema
* patient is between the ages of 1 month and 16 years
* accompanying adult is a primary caregiver
* child is not in foster care
* accompanying adult is 18 years old or older.

Exclusion Criteria:

* accompanying adult does not speak English
* accompanying adult is not the primary caregiver
* accompanying adult is not 18 years old or older
* patient is in foster care

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
change in eczema severity | 3 month follow-up
  eczema severity as measured by the Patient Oriented Eczema Measure (0-28 range, higher score=worse eczema severity)

SECONDARY OUTCOMES:
change in infant quality of life | 3 month follow-up
  infant quality of life as measured by the IDQOL (Infant's Dermatitis Quality of Life Index), uses a 0-30 scale, with a higher number reflecting worse quality of life. Used for children <4 years of age.
change in family quality of life | 3 month follow-up
  family quality of life as measured by the DFI (Dermatitis Family Impact Questionnaire), 0-30 scale with higher score reflecting worse quality of life
change in caregiver knowledge | 3 month follow-up
  change in caregiver knowledge pre-post as assessed by a questionnaire. This is not a standardized tool, but rather a series of 22 questions about caregiver comfort and understanding of eczema. Some responses use a likert scale format, while others are multiple choice questions. There are 8 multiple choice questions, each of which has one right answer. Those can be totaled to determine percentage correct.
change in child quality of life | 3 month follow-up
  child quality of life as measured by the CDLQI (Children's Dermatology Life Quality Index), uses a 0-30 scale, with a higher number reflecting worse quality of life. Used for children age 4-16.

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Rea, MD, MPH, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No